CLINICAL TRIAL: NCT02671383
Title: A Randomised, Open Label Switch Study Comparing Darunavir/Ritonavir 400mg/100mg Daily With Lopinavir/Ritonavir 800mg/200mg Daily, in HIV-positive Participants
Brief Title: Evaluation of Low-dose Darunavir in a Switch Study
Acronym: DRV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Willem Daniel Francois Venter (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor-Investigator, Willem Daniel Francois Venter, Professor, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRHI052
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: HIV Infections
Keywords: Antiretroviral Agents; Treatment; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darunavir (Active Comparator): Darunavir/Ritonavir 400/100mg once daily
  Interventions: Drug: Darunavir
- Lopinavir (Active Comparator): Lopinavir/Ritonavir 400/100mg twice daily
  Interventions: Drug: Lopinavir

INTERVENTIONS:
Drug: Darunavir — Darunavir/ritonavir 400/100mg (DRV/r) once daily plus nucleoside/nucleotide reverse transcriptase inhibitors.
  Other Names: Boosted darunavir (DRV/r)
  Arms: Darunavir
Drug: Lopinavir — Lopinavir/ritonavir 400/100mg (LPV/r) twice daily plus nucleoside/nucleotide reverse transcriptase inhibitors.
  Other Names: Boosted lopinavir (LVP/r)
  Arms: Lopinavir

SUMMARY:
This is a switch study to assess the non-inferiority (in terms of efficacy and safety) of darunavir (boosted with ritonavir, DRV/r 400mg/100mg daily) when compared with lopinavir (boosted with ritonavir, LPV/r total dose 800mg/200mg daily), in combination with a nucleoside backbone, administered as a second line therapy in HIV positive individuals.

DETAILED DESCRIPTION:
This is an open label randomised, parallel group, phase 3b, switch study to demonstrate non-inferiority of low-dose boosted darunavir (DRV/RTV 400/100 mg once daily) compared with boosted lopinavir-based (LPV/RTV 800/200 mg daily) second-line regimens when administered over 48 weeks in combination with two nucleos(t)ide reverse transcriptase inhibitors in patients infected with HIV-1 who are virologically suppressed and stable on a standard second-line regimen. All medications will be provided in an open-label design. Patients who are virologically suppressed and stable on a standard second-line regimen will be recruited for the study. There are concerns that switching these patients may result in virological failure as the study aimed at demonstrating non-inferiority of darunavir compared with Lopinavir. In such cases, the investigator will ensure that virological failures are investigated and patients are switched back to standard of care immediately. Participants will be patients who are receiving HIV treatment in public clinics. Interested patients will be invited to the study, information given, and only those who will give written informed consent will be screened, and if eligible enrolled into the study. Each enrolled participant will be follow-up at week 4, 12, 24, 36, and 48 (exit visit) from enrolment date. Data will be collected using ethics-approved worksheets, and captured into REDCap. The data manager will ensure data are correct and complete by performing data verifications - physical and electronic. Internal quality control will be performed by dedicated staff based on the study quality plan to be implemented. The external study monitor will perform 100% eligibility checks on all signed informed consents in addition to other source verifications during her periodic site visits according to the monitoring plan to be implemented. Findings from the monitor will be implemented in the form of data/procedure corrections per good clinical practice, and all relevant staff trained and documented accordingly. Participants' records will be coded and stored in a lockable cabinet. Only study staff will have access to participants' records. All electronic documents relating to the study will be stored in password-protected computers and only accessible to study staff. Study staff are not allowed to share password among themselves or with anyone outside the study team. Designed in non-inferiority fashion, this study will enrol approximately 300 participants for 80% power to detect a 10% non-inferiority margin in the per protocol (PP) analysis. A Data Safety Management Board (DSMB) will oversee and review the interim data report. At the close of the study, results will be disseminated to participants, and the scientific community, as well as updated on clinicaltrial.gov.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥18 years
* Participant weight >40kg
* Participant is on a LPV/r-containing regimen for at least 6 months with no history of other protease inhibitors
* Participant has a plasma HIV-1 RNA level <50 copies/mL in the last 60 days
* Participant is informed and has the ability to comprehend the full nature and purpose of the study, and give voluntary written informed consent before inclusion in the study

Exclusion Criteria:

* Participants who are taking any antiretrovirals other than nucleoside/nucleotide reverse transcriptase inhibitors and LPV/r
* Any prior history of genotype-documented protease inhibitor resistance
* Participants who are taking rifampicin or any other therapy with major cytochrome P450 interactions, within the last month
* Participants who are allergic to sulphonamides
* Participants who have a current history of drug or alcohol abuse that, in the opinion of the investigator, may be an impediment to participant adherence to the protocol
* Female participants who are currently pregnant or breastfeeding
* Female participants desiring pregnancy during the next year
* Participants who have a strong likelihood of relocating far enough to make access to the study site difficult
* Any condition(s) or laboratory report that, in the opinion of the investigator, might put the participant at risk, or interfere with the study objectives or the participant's adherence to study requirements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with undetectable HIV-1 RNA levels | Week 48
Number of participants with certain adverse events related to the treatment | Week 48

SECONDARY OUTCOMES:
Time to virologic failure | Week 48

OTHER OUTCOMES:
Lipids measure | Baseline, Week 24 and 48
Fasting glucose measure | Baseline and Week 48
Creatinine clearance measure | Baseline, Week 12, 24, and 48

CONTACTS AND LOCATIONS:
Locations (1):
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Draaijer M, Lalla-Edward ST, Venter WDF, Vos A. Phone Calls to Retain Research Participants and Determinants of Reachability in an African Setting: Observational Study. JMIR Form Res. 2020 Sep 30;4(9):e19138. doi: 10.2196/19138. PMID 32996891
- [Derived] Venter WDF, Moorhouse M, Sokhela S, Serenata C, Akpomiemie G, Qavi A, Mashabane N, Arulappan N, Sim JW, Sinxadi PZ, Wiesner L, Maharaj E, Wallis C, Boyles T, Ripin D, Stacey S, Chitauri G, Hill A. Low-dose ritonavir-boosted darunavir once daily versus ritonavir-boosted lopinavir for participants with less than 50 HIV RNA copies per mL (WRHI 052): a randomised, open-label, phase 3, non-inferiority trial. Lancet HIV. 2019 Jul;6(7):e428-e437. doi: 10.1016/S2352-3018(19)30081-5. Epub 2019 Jun 12. PMID 31202690